CLINICAL TRIAL: NCT05383443
Title: Multiple Interventions to Prevent Cognitive Decline (MIND-Matosinhos) - a Randomized Controlled Trial
Brief Title: MIND-Matosinhos: Multiple Interventions to Prevent Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Saude Publica da Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 63/CE/JAS/2020
Record Dates: First submitted 2022-05-03; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Cognitive Dysfunction; Cognition Disorder; Memory Disorders; Cognitive Impairment; Neurocognitive Disorders
Keywords: Aging; Cognitive Dysfunction; Cognition Disorders; Dementia; Diet, Healthy; Exercise Therapy; Hearing Loss; Memory Disorders; Multidomain intervention; Randomized Controlled Trial
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders; Memory Disorders; Neurocognitive Disorders; Dementia; Hearing Loss | interventions — Cognitive Training; Exercise; Nutrition Assessment; Correction of Hearing Impairment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Multidomain non-pharmacological intervention, including cognitive training, physical exercise, nutrition education, capacitation to deal with cognitive decline, and diagnosis and correction of hearing impairment.
  The intervention plan includes home training activities of identical intensity for participants with and without access or autonomy to use computer/internet. It will comprise individual and group sessions over three months, possibly extensible up to 12 months.
  Caregivers or partners of all participants will be invited to participate in the activities of nutrition education and capacitation to deal with cognitive decline.
  Interventions: Behavioral: Cognitive training; Behavioral: Physical exercise; Behavioral: Nutrition education; Behavioral: Capacitation to deal with cognitive decline; Other: Diagnosis and correction of hearing impairment
- Control group (Active Comparator): Multidomain non-pharmacological intervention, including cognitive training, physical exercise, nutrition education, capacitation to deal with cognitive decline, and diagnosis and correction of hearing impairment.
  It will comprise individual and group sessions, over three months (possibly extensible up to 12 months), conducted with a lower frequency in comparison with the intervention group.
  Caregivers or partners of all participants will be invited to participate in the activities of nutrition education and capacitation to deal with cognitive decline.
  Interventions: Behavioral: Cognitive training; Behavioral: Physical exercise; Behavioral: Nutrition education; Behavioral: Capacitation to deal with cognitive decline; Behavioral: Diagnosis and correction of hearing impairment

INTERVENTIONS:
Behavioral: Cognitive training — This component will comprise the following activities:
  i. In-person group training (monthly): 60-minute sessions, supervised by a psychologist; ii. Home individual training (≥5 times per week): unsupervised 30-minutes remote sessions, using the COGWEB® online platform or paper/pencil exercises (for those participants without computer/internet or who do not use one autonomously).
  Arms: Intervention
Behavioral: Physical exercise — This component will be based on 60-minute sessions including aerobic, resistance, agility/balance and flexibility exercises, supervised by a physical education teacher:
  i. In-person group training (monthly); ii. In-person group training or remote synchronous training (group) or provision of education booklets with photos and exercise instructions to be performed individually (twice weekly), depending on the evolution of the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) pandemic.
  Arms: Intervention
Behavioral: Nutrition education — This component will be based on the following activities:
  i. In-person group 120-minute sessions (monthly), guided by a nutritionist, comprising: presentation and discussion of healthy and easy to cook recipes by the nutritionist and preparation of healthy meals by the participants; ii. In-person individual appointment with a nutritionist (monthly).
  Arms: Intervention
Behavioral: Capacitation to deal with cognitive decline — This component will be based on in-person 60-minute group sessions (monthly), guided by a psychologist, allowing participants to share experiences and learn strategies to cope with cognitive decline in their daily life.
  Arms: Intervention
Other: Diagnosis and correction of hearing impairment — This component will be based on an evaluation session conducted by otolaryngologists and audiologists, who will evaluate previous hearing problems and use of hearing aids, and will include an otoscopy and an audiogram.
  Arms: Intervention
Behavioral: Cognitive training — This component will comprise the following activities:
  i. In-person group training (monthly): 60-minute sessions, supervised by a psychologist; ii. Home individual training (once a week): unsupervised 30-minutes remote sessions, using the COGWEB® online platform or paper/pencil exercises (for those participants without computer/internet or who do not use one autonomously).
  Arms: Control group
Behavioral: Physical exercise — In-person group training (monthly): 60-minute sessions including aerobic, resistance, agility/balance and flexibility exercises, supervised by a physical education teacher.
  Arms: Control group
Behavioral: Nutrition education — In-person group 120-minute sessions (monthly), guided by a nutritionist, comprising: presentation and discussion of healthy and easy to cook recipes by the nutritionist and preparation of healthy meals by the participants. The participants will have the opportunity to consume the prepared meals at home.
  Arms: Control group
Behavioral: Capacitation to deal with cognitive decline — In-person group 60-minute sessions (monthly), guided by a psychologist, allowing participants to share experiences and learn strategies to cope with cognitive decline in their daily life.
  Arms: Control group
Behavioral: Diagnosis and correction of hearing impairment — This component will be based on an evaluation session conducted by otolaryngologists and audiologists, who will evaluate previous hearing problems and use of hearing aids, and will include an otoscopy and an audiogram.
  Arms: Control group

SUMMARY:
The present study aims to quantify the impact of a multidomain approach to prevent cognitive decline in individuals from the general population at-high risk of dementia. It will be based on five distinct components: 1) cognitive training; 2) physical exercise; 3) nutrition education; 4) capacitation to deal with cognitive decline; 5) assessment and correction of hearing loss.

DETAILED DESCRIPTION:
This is a community-based randomized controlled trial (RCT), which will be implemented in Matosinhos municipality (Portugal) and will be conducted over three months, possibly extensible up to 12 months.

Eligible individuals (n=300) will be randomized (1:1) into two arms: intervention and control groups. The intervention plan will be composed by five non-pharmacological strategies, namely: 1) cognitive training; 2) physical exercise; 3) nutrition education; 4) capacitation to deal with cognitive decline; 5) assessment and correction of hearing loss. This plan will be applied to both groups, but with lower intensity among the control group.

Participants' characteristics will be assessed at baseline and at three months; for those who complete one year of intervention, additional follow-ups at six and 12 months after the beginning of the intervention will be conducted. These evaluations will cover the following domains: sociodemographic, lifestyle, health and anthropometric characteristics; cognitive function; subjective memory complains; symptoms of anxiety and depression; quality of life; physical performance; levels of glycated hemoglobin and 24-hour urinary sodium, potassium, creatinine excretion as well as pH.

The results of the present study may guide future clinical practices and health policies aiming to prevent cognitive decline and reduce the overall burden of dementia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years;
* Score equal or higher than the validated cutoff points defined as 2 standard deviations below the mean for age and education in the Montreal Cognitive Assessment (MoCA);
* ≥6 points on the Cardiovascular Risk Factors, Aging and Dementia Dementia Risk Score (CAIDE);
* ≥4 years of schooling.

Exclusion Criteria:

* Medical disability that contraindicates physical activity;
* Lack of autonomy in daily activities;
* Previous diagnosis of dementia or severe incapacity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet | Up to 12 months
  Variation of participant's self-reported adherence to the Mediterranean diet, assessed using the Mediterranean food pattern scale (MEDAS), between the baseline assessment and the end of follow-up. This scale varies from 0 (lowest adherence to the Mediterranean diet) to 14 points (highest adherence to the Mediterranean diet). A score over 10 points indicates good adherence to the Mediterranean diet.
Self-reported quality of life | Up to 12 months
  Variation of participant's quality of life, assessed using the EuroQol Group scale - 5 dimensions (EQ-5D) scale, between the baseline assessment and the end of follow-up. This scale is subdivided in two subscales: a) five multiple choice questions, with five response possibilities, which produce a score that varies from 5 (best score) to 25 points (worst score); b) visual analogic scale, that varies from 0 (worst score) to 100 (best score).

SECONDARY OUTCOMES:
Memory complaints | Up to 12 months
  Variation of the self-reported memory complaints, assessed using the Subjective Memory Complaints Scale, between the baseline assessment and the end of follow-up. This scale varies from 0 (best score) to 21 points (worst score). Scores over three points indicate the presence of self-reported memory complaints.
Cognitive performance 1 | Up to 12 months
  Variation of participant's cognitive performance assessed using the Montreal Cognitive Assessment, between the baseline assessment and the end of the follow-up. This scale varies from 0 (worst cognitive performance) to 30 points (best cognitive performance).
Cognitive performance 2 | Up to 12 months
  Variation of participant's cognitive performance assessed using a neuropsychological battery tests, between the baseline assessment and the end of the follow-up. This will be reported in the format of a Z-score, assuming positive and negative values. Higher scores indicate better cognitive performance.
Anxiety and depression | Up to 12 months
  Variation of the anxiety and depression scores, assessed using the Hospital Anxiety and Depression Scale (HADS), between the baseline assessment and the end of the follow-up. This scale varies from 0 (best score) to 21 points (worst score).
Handgrip strength | Up to 12 months
  Variation of participant's handgrip strength, assessed using a dynamometer, between the baseline assessment and the end of the follow-up.
Agility 1 | Up to 12 months
  Variation of participant's agility and balance, assessed using the Timed Up and Go Test scale, between the baseline assessment and the end of the follow-up. This is measured in time units (seconds) and varies from 0 (best score) to infinite (worst score).
Agility 2 | Up to 12 months
  Variation of participant's agility and balance, assessed using the Unipedal Stance Test, between the baseline assessment and the end of the follow-up. This is measured in time units (seconds) and varies from 0 (best score) to infinite (worst score).
Upper body strength | Up to 12 months
  Variation of participant's upper body strength assessed using the 30-second arm curl test from the Senior Fitness Test.
Lower body strength | Up to 12 months
  Variation of participant's lower body strength assessed using the 30-second chair stand test from the Senior Fitness Test.
Upper body flexibility | Up to 12 months
  Variation of participant's upper body flexibility assessed using the back-scratch test from the Senior Fitness Test.
Lower body flexibility | Up to 12 months
  Variation of participant's lower body flexibility assessed using the chair sit-and-reach test from the Senior Fitness Test.
Agility 3 | Up to 12 months
  Variation of participant's agility and dynamic balance assessed using the 8-foot distance test (2,44 meters) from the Senior Fitness Test.
Aerobic endurance | Up to 12 months
  Variation of participant's aerobic endurance assessed using the 2-minute step test from the Senior Fitness Test.
Lower limb function | Up to 12 months
  Variation of participant's lower limb function, assessed using the Short Physical Performance Battery (SPPB), which tests 3 dimensions: standing balance, walking speed, and chair stands. Each component is scored between 0-4; total score ranges from 0 (poor performance) to 12 (best performance).
Levels of glycated hemoglobin | Up to 12 months
  Variation of participant's levels of glycated hemoglobin, between the baseline assessment and the end of follow-up. This parameter will be measured through a laboratory analysis of participants' blood sample and will be used to analyze glycemic control.
24-hour urinary sodium excretion | Up to 12 months
  Variation of participant's urinary sodium excretion, between the baseline and the follow-up assessments. This parameter will be measured through a laboratory analysis of participants' 24-hour urinary samples and will be analyzed as a proxy of dietary salt intake.
24-hour urinary potassium excretion | Up to 12 months
  Variation of participant's urinary potassium excretion, between the baseline and the follow-up assessments. This parameter will be measured through a laboratory analysis of participants' 24-hour urinary samples and will be analyzed as a proxy of dietary potassium intake.
Body mass index | Up to 12 months
  Variation of participant's body mass index between the baseline assessment and the end of follow-up.
Blood pressure | Up to 12 months
  Variation of participant's systolic and diastolic blood pressure, between the baseline evaluation and the end of follow-up.
Functional capacity to perform instrumental activities of daily living | Up to 12 months
  Variation of participant's independence on performing instrumental activities of daily living, using the Lawton & Brody scale, which ranges from 0 to 8 and higher scores represent increased functional capacity to perform instrumental activities.
Time of follow-up | Up to 12 months
  Number of days between the first and the last session attended by the participant.
Implemented sessions | Up to 12 months
  Proportion of sessions implemented, calculated as the number of sessions that the research team was able to implement divided by the total number of sessions planned.
Complete assessment of participants | Up to 12 months
  For each study outcome, proportion of participants with complete information, calculated at baseline and different moments of follow-up, as the number of participants with complete information divided by the total number of participants evaluated.
Adherence to each component of the intervention | Up to 12 months
  Proportion of adherence to each component of the intervention and to different intervention modalities (remote/in person), calculated as the number of sessions attended divided by the total number of sessions implemented. For remote cognitive training the outcome will be the absolute number of sessions.
Dropout | Up to 12 months
  Proportion of participants who dropped out of the study, calculated as the number of participants who dropped out after attending at least one session divided by the total number of participants who attended at least one session.

CONTACTS AND LOCATIONS:
Overall Officials: Vítor Tedim Cruz, PhD, Principal Investigator — Instituto de Saude Publica da Universidade do Porto
Locations (1):
- Instituto de Saúde Pública da Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No